CLINICAL TRIAL: NCT03800498
Title: Shalamar Institute of Health Sciences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Open University Islamabad (Other)
Responsible Party: Principal Investigator, Naiza Yousef, Student, Allama Iqbal Open University Islamabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIHS
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Effect of Didactic Intervention Regarding (DASH) on Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): For twelve weeks, only intervention group were given DASH education
  Interventions: Other: DASH Education
- Controlled (No Intervention): Controlled group not received DASH education

INTERVENTIONS:
Other: DASH Education — DASH health education about general knowledge of DASH diet Plan and lifestyle modification
  Arms: Intervention

SUMMARY:
Effect of Didactic intervention regarding Dietary Approach to Stop Hypertension (DASH) on Hypertensive Patients Blood Pressure, Knowledge and Attitude at a Tertiary Hospital of Lahore

DETAILED DESCRIPTION:
Objective: To explore the effect of didactic intervention regarding dietary approach to stop hypertension (DASH) on hypertensive patients blood pressure, knowledge and attitude.

Study Design: Randomized controlled trial Place and Duration of Study: Punjab Institute of Cardiology (PIC) Lahore. From June 2018 to Oct 2018.

Methodology: Seventy volunteers aged 20-60 years attending regularly outpatient department at Punjab institute of cardiology Lahore, with systolic > 130 mm hg, diastolic > 80 mm hg were selected and assigned into 2 groups, i.e. Intervention and control, by simple random lottery method. For twelve weeks, only intervention group were given DASH education. Both groups were checked for DASH knowledge, attitude, and systolic diastolic blood pressure, before and after education session. Pre-tested questionnaire was used for demographic, attitude and knowledge data collection.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patient aged 20-60 years attending regularly at Punjab institute of cardiology outpatient department Lahore
* systolic > 130 mm hg
* diastolic > 80 mm hg.

Exclusion Criteria:

* Less than 20 years age
* patient diagnosed with secondary hypertension
* any mental and physical ailment that may interfere the intervention like deafness and blindness.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Pre-tested questionnaire was used | 1 month
  10 knowledge questions were asked with minimum score 0 and maximum 10. Attitude assessment consisted of 4 questions and score range was 0-4.

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Ahmad, PhD, Principal Investigator — Shalamar Institute of Health Sciences
Locations (1):
- Nazia, Lahore, Punjab Province, Pakistan